CLINICAL TRIAL: NCT05997043
Title: Safety and Efficacy of Botulinum Toxin A for Treatment of Overactive Bladder in Parkinson's Disease:Randomized Controlled Trial
Brief Title: Safety and Efficacy of Botulinum Toxin A for Treatment of Overactive Bladder in Parkinson's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Shuzhen Zhu, Deputy Chief Physician, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-KY-301-02
Record Dates: First submitted 2023-08-06; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Parkinson's Disease; Overactive Bladder; Onabotulinumtoxin A
MeSH Terms: conditions — Parkinson Disease; Urinary Bladder, Overactive | interventions — Antiparkinson Agents

STUDY DESIGN:
Intervention Model Description: The intervention group was given oral anti-Parkinson's drugs and Botox injection, while the control group was given only anti-Parkinson's drugs.
Who Masked: Outcomes Assessor
Masking Description: For Parkinson's disease patients with overactive bladder, participants were assigned to an experimental or control group in a 1:1 ratio at the end of the baseline visit.Assignment will be concealed (sealed envelopes) and randomized to either the experimental or control group using an independent online computerized randomization system. Once randomized into the study, all patients will be included in the ITT analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group
  Interventions: Drug: oral anti-Parkinson drugs and injection of botulinum toxin
- Control group (Placebo Comparator): Control group
  Interventions: Drug: oral anti-Parkinson's drugs

INTERVENTIONS:
Drug: oral anti-Parkinson drugs and injection of botulinum toxin — The experimental group was treated with oral anti-Parkinson drugs and injection of botulinum toxin
  Arms: Experimental group
Drug: oral anti-Parkinson's drugs — The control group only took oral anti-Parkinson's drugs.
  Arms: Control group

SUMMARY:
A randomized controlled trial is to be conducted to confirm the efficacy and safety of intramuscular injection of botulinum toxin in the treatment of Parkinson's bladder overactivity.

DETAILED DESCRIPTION:
Overactive bladder is defined by the International Continence Society as a syndrome characterized by symptoms of urinary urgency, often accompanied by frequency and nocturia, with or without urge incontinence, but without urinary tract infection or other definite symptoms pathological changes.

Bladder dysfunction is one of the most common autonomic nervous disorders in Parkinson's disease (PD). Up to 70% of PD patients have bladder hyperactivity. Nocturia is the most commonly reported symptom , followed by urinary frequency, urinary urgency and urge incontinence, affecting patients' quality of life and social life.

At present, intramuscular injection of 100U botulinum toxin (BoNT-A) is a reasonable choice for the treatment of bladder overactivity in PD, and it has been proved to be a safe and effective method for the treatment of neurogenic detrusor overactivity, especially for patients with insufficient response to anticholinergic drugs,which is a Grade Ia recommendation in the EAU guidelines.

There are some problems in the current research as follows: 1. Single-arm study, non-randomized control, and small sample size; 2. Only patients with urinary incontinence but not patients with dry bladder overactivity were included; 3. Patients with urinary retention are not excluded, resulting in urinary retention after injection of botulinum toxin, affecting the experience of patients; 4. Botulinum toxin dose injection varies, there is still a lack of large-scale prospective clinical studies to reflect the relationship between botulinum toxin dose and residual urine volume; 5. The urodynamic index was used in the outcome index, which could not reflect the improvement of symptoms sensitively and objectively. In order to make up for the shortcomings of previous studies, a randomized controlled trial is planned to confirm the efficacy and safety of intramuscular injection of low dose botulinum toxin in the treatment of PD bladder overactivity

ELIGIBILITY:
Inclusion Criteria:

1. patients with idiopathic Parkinson's disease were diagnosed by experienced neurologists based on the diagnostic criteria of the International Motor Disorder Association.
2. PD patients with overactive bladder were observed by voiding diary for 3 days and evaluated by OABSS score.
3. Eligible males and females, aged between 25 and 80.
4. The patient was treated with dopaminergic drugs, and if there was an wearing-off phenomenon, it was evaluated during the turning-off period or without taking the drug (when the patient developed one of the symptoms in WOQ-19 [13] and the symptom improved after the next medication, it suggested that there was an end-of-dose phenomenon).
5. With a history of NDO ≥ 3 months, the symptoms of bladder overactivity were not fully controlled by anticholinergic drugs, which was defined as insufficient response after 4 weeks of treatment or unbearable side effects after 2 weeks of optimized dose treatment.
6. patients who took anticholinergic drugs at baseline must maintain a stable dose throughout the study, while those who did not take anticholinergic drugs could not take them during the study period.
7. if necessary, the patient must be willing to initiate intermittent catheterization (CIC).
8. the informed consent of the subject or his guardian has been obtained, and the informed consent of the clinical trial has been signed voluntarily.

Exclusion Criteria:

1) Ultrasonography showed that the residual urine of bladder was larger than 10ml. 2) Patients with glaucoma and myasthenia gravis are not suitable for botulinum toxin.

3) Indwelling catheter or intermittent catheterization (CIC) is needed to empty the bladder.

4) Patients have been treated with botulinum toxin for any urinary disease. 5) People who are known to be allergic or allergic to drugs and their ingredients 6) Take drugs that interfere with neuromuscular transmission. 7) Receiving anticoagulant therapy. 8) There is infection at the injection site. 9)With dementia, Parkinson's dementia scale ≤ 73.5 at screening time [15] or with Parkinson's disease psychiatric disorder

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-26 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Symptom score of overactive bladder | 2 weeks,1month,2 month, 3 month
  The purpose of this questionnaire is to assess the severity of symptoms in patients with overactive bladder. Based on the OABSS scale, when the score of question 3 (urgency) is more than 2 points, and the whole OABSS score is more than 3 points, it can be diagnosed as OAB

SECONDARY OUTCOMES:
urinary symptoms | 2 weeks,1month,2 month, 3 month
  frequency、urgency、noturia and urge incontinence
urodynamics | 2 weeks,1month,2 month, 3 month
  first sensation、first desire to void、strong desire to void、maximum bladder capacity
King health score | 2 weeks,1month,2 month, 3 month
  This questionnaire contains 9 areas, of which the general perception of health (GHP) and the severity of urination problems (SUP) contain only one problem, and the other 7 areas each contain multiple problems. The seven areas were behavioral limitation (RL), social limitation (SL), movement limitation (PL), personal life (PR), emotion (EMO), sleep / energy (SE) and urinary incontinence coping style (CM).
Urgency severity scale | 2 weeks,1month,2 month, 3 month
  This questionnaire evaluates the degree of urination urgency. It is divided into 5 grades from 0 to 4, which are no sense of urgency, slight sense of urgency, moderate urgency, severe urgency and leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhen Zhu, Doctor, Study Director — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China